CLINICAL TRIAL: NCT04153344
Title: Function of the Pigment Epithelium in Patients With Type 1 Neurofibromatosis
Acronym: NEF-1
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190937; 2019-A02526-51 (Other: ID RCB)
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Neurofibromatosis Type 1
Keywords: Neurofibromatosis type 1; Infrared hyperreflective areas; Hyperactivity of the pigment epithelium; Electro-oculogram; Electroretinogram
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Infrared hyperreflective area: Patients with neurofibromatosis type 1 and with infrared hyperreflective areas
  Interventions: Other: Electro-oculogram; Other: Full-field electroretinogram
- No infrared hyperreflective areas: Patients with neurofibromatosis type 1 and with no infrared hyperreflective areas
  Interventions: Other: Electro-oculogram; Other: Full-field electroretinogram
- Controls: Patients with no neurofibromatosis type 1
  Interventions: Other: Electro-oculogram; Other: Full-field electroretinogram

INTERVENTIONS:
Other: Electro-oculogram — Electrophysiological recording of changes in electrical potential across the retinal pigmentary epithelium during successive periods of dark and light adaptation, according to ISCEV standards. Results will comprise dark trough value and light/dark (Arden) ratio.
Other: Full-field electroretinogram — Electrophysiological recording of retinal function. Results will comprise amplitudes and latencies of each electroretinography response (dark-adapted 0.01, dark-adapted 3.0, dark-adapted 10.0, dark-adapted 3.0 oscillatory potentials, light-adapted 3.0, light-adapted 3.0 flicker).

SUMMARY:
The objective of this study is to study the function of the pigment epithelium in patients with neurofibromatosis type 1 using electro-oculogram to confirm abnormally high values reported in previous studies, but also to correlate this hyperactivity of the pigment epithelium with the presence and size of choroidal hyperreflective areas observed in infra-red imaging of the fundus.

The hypothesis of the study is that the function of the pigment epithelium measured by the electro-oculogram correlates with the surface of choroidal hyperreflective areas. Finally, the potential consequences of a supra-normal function of the pigment epithelium on the global retinal function are not known. A full-field electroretinogram will evaluate the global neurosensory retinal function.

DETAILED DESCRIPTION:
Patients with neurofibromatosis type 1 have numerous eye problems: glioma of the optic pathways, Lisch nodules, palpebral involvement by plexiform neurofibromas, orbital dysplasia, etc. With the emergence of multimodal imaging in ophthalmology a new ocular involvement has been described: choroidal hyperreflective areas. They are located in the most superficial layers of the choroid, adjacent to the retinal pigment epithelium, visible only on infra-red imaging of the fundus. These areas are frequently observed, about 90% in adults and 70 to 80% in children. With a sensitivity of 0.83 and a specificity of 0.96, these lesions would have their place as a diagnostic criterion for neurofibromatosis type 1.

In parallel, two successive studies have evaluated the function of the retinal pigment epithelium using electro-oculograms; they showed in patients with neurofibromatosis type 1 a significant increase in the Arden ratio, reflecting hyperactivity of the pigment epithelium.

The objective of this study is to study the function of the pigment epithelium in patients with neurofibromatosis type 1, using electro-oculogram to confirm these abnormally high values, but also to correlate this hyperactivity of the pigment epithelium to the presence and total area of choroidal lesions observed in infra-red imaging of the fundus.

The hypothesis of the study is that the function of the pigment epithelium measured by the electro-oculogram correlates with the surface of the choroidal hyperreflective areas. Finally, the potential consequences of a supra-normal function of the pigment epithelium on the global retinal function are not known. A full-field electroretinogram will evaluate the global neurosensory retinal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neurofibromatosis type 1, aged 7 years or older:

  * Presence of hyper-reflective choroidal lesions in infra-red imaging in the group with choroidal lesions.
  * Absence of hyper-reflective choroidal lesions in infra-red imaging in the group without choroidal lesions.
* Control patients free from retinal or choroidal pathology, matched for age to patients in the group with neurofibromatosis type 1.
* Patients consulting the ophthalmology department of Necker-Enfants Malades Hospital.
* Non-opposition of the holders of the parental authority and the minor patient; non-opposition of the major patient.

Exclusion Criteria:

* Impossibility to perform an electro-oculogram, especially because of an oculomotor disorder, or an electroretinogram, for example because of hyperactivity.
* Significant impairment of visual function.
* Retinal pathology proved.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients consulting the ophthalmology department of Necker-Enfants Malades Hospital:
  * 10 patients with neurofibromatosis type 1 without infrared hyperreflective areas
  * 10 patients with neurofibromatosis type 1 and infrared hyperreflective areas
  * 10 control patients with no retinal disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Dark trough value | 12 months
  Electro-oculogram : dark trough value (μV).
Light/dark (Arden) ratio | 12 months
  Electro-oculogram : ratio between the light and dark potentials.

SECONDARY OUTCOMES:
Number and area of infrared hyperreflective areas | 12 months
  Infrared fundus picture.
Values of the amplitudes | 12 months
  Electroretinogram : values of the amplitudes (μV) of a- and/or b-waves for dark-adapted 0.01, dark adapted 3.0, dark-adapted 10.0, dark-adapted 3.0 oscillatory potentials, light-adapted 3.0, and light-adapted 3.0 flicker.
Values of the peak times | 12 months
  Electroretinogram : values of the peak times (ms) of a- and/or b-waves for dark-adapted 0.01, dark adapted 3.0, dark-adapted 10.0, dark-adapted 3.0 oscillatory potentials, light-adapted 3.0, and value of the peak-to-peak time (ms) for light-adapted 3.0 flicker.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Robert, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Dominique Brémond-Gignac, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lubinski W, Zajaczek S, Sych Z, Penkala K, Palacz O, Lubinski J. Electro-oculogram in patients with neurofibromatosis type 1. Doc Ophthalmol. 2001 Sep;103(2):91-103. doi: 10.1023/a:1012271206258. PMID 11720259
- [Background] Viola F, Villani E, Natacci F, Selicorni A, Melloni G, Vezzola D, Barteselli G, Mapelli C, Pirondini C, Ratiglia R. Choroidal abnormalities detected by near-infrared reflectance imaging as a new diagnostic criterion for neurofibromatosis 1. Ophthalmology. 2012 Feb;119(2):369-75. doi: 10.1016/j.ophtha.2011.07.046. Epub 2011 Oct 2. PMID 21963267
- [Background] Touze R, Abitbol MM, Bremond-Gignac D, Robert MP. Function of the Retinal Pigment Epithelium in Patients With Neurofibromatosis Type 1. Invest Ophthalmol Vis Sci. 2022 Apr 1;63(4):6. doi: 10.1167/iovs.63.4.6. PMID 35394491